CLINICAL TRIAL: NCT05486325
Title: Pilot Study of the Endolumik Gastric Calibration Tube for Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Endolumik, Inc (Industry)
Collaborators: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00058006
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: The sample size (n) will be 20-30 Bariatric patients. Twenty participants will undergo laparoscopic or robotic sleeve gastrectomy using the Endolumik Gastric Calibration Tube instead of the standard bougie calibration tube.
  Ten participants will undergo laparoscopic gastric bypass using the Endolumik Gastric Calibration Tube instead of the standard calibration tube.
  The current pilot protocol is a qualitative, not quantitative, study design, thus no power calculation is indicated. The goal of the present pilot study is to serve as the First In Human trial and confirm that the Endolumik Gastric Calibration Tube performs similar to predicate devices currently on the market, as well as to get end-user feedback prior to 510(k) application to the FDA. The sample size was chosen because 20 to 30 uses will allow the development team to appropriately evaluate device performance.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Bariatric Surgery (Experimental): Up to twenty participants meeting inclusion criteria will undergo laparoscopic or robotic sleeve gastrectomy using the Endolumik Gastric Calibration Tube instead of the standard bougie calibration tube. Up to ten participants meeting inclusion criteria will undergo laparoscopic gastric bypass using the Endolumik Gastric Calibration Tube instead of the standard calibration tube.
  Interventions: Device: Endolumik Gastric Calibration Tube (EGCT)

INTERVENTIONS:
Device: Endolumik Gastric Calibration Tube (EGCT) — Up to twenty participants will undergo laparoscopic or robotic sleeve gastrectomy using the EGCT. This operation will take approximately 60 minutes.
  The portions of the sleeve gastrectomy operation where the EGCT will be used include:
  * To evacuate gastric contents
  * During construction of the gastric sleeve
  * To perform the leak test of the gastric sleeve Up to ten participants will undergo laparoscopic gastric bypass using the EGCT. This operation will take approximately 120 minutes.
  The portions of the gastric bypass operation where the EGCT will be used include:
  * To evacuate gastric contents
  * During construction of the gastric pouch
  * To calibrate closure of the gastrojejunal anastomosis
  * To perform a leak test of the gastrojejunal anastomosis In both procedures, The amount of time the EGCT will be inside the patient is approximately 20 minutes. The device is removed prior to the conclusion of the operation, while the patient is under anesthesia.

SUMMARY:
The pilot study will be a First In Human Clinical Trial to evaluate the Endolumik Gastric Calibration Tube and associated methods in a human clinical cohort of 20-30 bariatric patients at two high-volume bariatric programs. During this clinical study, the single-use, disposable Endolumik Gastric Calibration Tube will be used during twenty sleeve gastrectomy operations and gastric bypass operations.

DETAILED DESCRIPTION:
Endolumik Inc. has developed a fluorescence-guided calibration device, the Endolumik Gastric Calibration Tube, to improve visualization during bariatric operations. The present pilot study will be a First In Human Clinical Trial to evaluate the Endolumik Gastric Calibration Tube and associated methods in a human clinical cohort of 20-30 bariatric patients at two high-volume bariatric programs. During this clinical study, the single-use, disposable Endolumik Gastric Calibration Tube will be used during twenty sleeve gastrectomy operations and gastric bypass operations. The goal of the present study is to confirm that the Endolumik Gastric Calibration Tube performs similar to predicate devices currently on the market, as well as to get end-user feedback prior to submitting a 510(k) application to the U.S. Food and Drug Administration (FDA).

In this multicenter trial, both study sites are certified as Bariatric Centers of Excellence through the American Society of Metabolic and Bariatric Surgery. The first clinical site is Ruby Memorial Hospital, part of West Virginia University; the second clinical site is Durham Regional Hospital, part of Duke University.

To date, using funding from a West Virginia Clinical & Translational Science Institute Launch Pilot Grant, our team has validated the device and associated methods of fluorescence-guided sleeve gastrectomy and fluorescence-guided gastric bypass in ex-vivo and in-vivo porcine models, as well as human cadaveric tissue models. Based on FDA criteria, this investigational device meets the definition of a Non-Significant Risk (NSR) device; the risk classification document is included with submission materials.

The investigational device provided will have met design controls per FDA code of federal regulation (CFR): 21 CFR 820.30. Endolumik Inc. will serve as the industry sponsor for this study and will donate the devices being used for the protocol to the two participating study sites. Development of the technology in this research is supported by the West Virginia University Department of Surgery.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Adults (between age of 18 and 65 years old)
* Have body mass index (BMI) between 35 and 65.99 kg/m2
* Male or female bariatric patients undergoing bariatric surgery at one of the two sites included in the protocol.

Exclusion Criteria:

* Nonbariatric patients
* Patients who have conditions that preclude a sleeve gastrectomy or gastric bypass operation
* Patients with esophageal stricture
* Patients with esophageal varices
* Patients with a Zenker's diverticulum
* Patients aged 66 and older
* Patients with a BMI of 66 kg/m2 or greater
* Pregnant Women
* Lactating Women
* Other vulnerable patient populations: pregnant and lactating women, prisoners, cognitively impaired and critically ill subjects.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Intraoperative adverse events | During surgical treatment
  Adverse events occurring during surgical treatment
Operative time | During surgical treatment
  Duration of surgical treatment
30-day morbidity | 30 days post surgical treatment
  any 30-day Metabolic and Bariatric Surgery Accreditation and Quality Improvement Program (MBSAQIP) Occurrences

CONTACTS AND LOCATIONS:
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] English WJ, DeMaria EJ, Brethauer SA, Mattar SG, Rosenthal RJ, Morton JM. American Society for Metabolic and Bariatric Surgery estimation of metabolic and bariatric procedures performed in the United States in 2016. Surg Obes Relat Dis. 2018 Mar;14(3):259-263. doi: 10.1016/j.soard.2017.12.013. Epub 2017 Dec 16. PMID 29370995
- [Background] Mahawar KK. Bougie-Related Oesophageal Injury with Bariatric Surgery: An Unrecognised Problem. Obes Surg. 2016 Aug;26(8):1935-6. doi: 10.1007/s11695-016-2213-1. No abstract available. PMID 27129804
- [Background] Lovece A, Rouvelas I, Hayami M, Lindblad M, Tsekrekos A. Cervical esophageal perforation caused by the use of bougie during laparoscopic sleeve gastrectomy: a case report and review of the literature. BMC Surg. 2020 Jan 10;20(1):9. doi: 10.1186/s12893-020-0679-1. PMID 31924187
- See also: Morbid Obesity Data — https://www.who.int/news-room/fact-sheets/detail/obesity-and-overweight
- See also: Bariatric Surgery Data — https://asmbs.org/resources/estimate-of-bariatric-surgery-numbers
- See also: Fluorescence Guided Surgery — https://pubmed.ncbi.nlm.nih.gov/?term=fluorescence+guided+and+surgery+or+indocyanine+green+and+surgery

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT05486325/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/25/NCT05486325/ICF_001.pdf